CLINICAL TRIAL: NCT00818025
Title: Phase III Trial of Pocket PATH: A Computerized Intervention to Promote Self-Care
Brief Title: Comparing Methods for Tracking Health Information at Home After Lung Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Annette DeVito Dabbs, PhD, RN, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO08070401; 1R01NR010711-01 (NIH)
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Lung Disease
Keywords: Transplantation; Self-care agency; Self-care behaviors; Hand-held device
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention): All subjects will receive standard care to prepare for discharge that consists of a one-on-one, pre-discharge educational session delivered by the transplant coordinator prior to hospital discharge and provision of a reference binder for each lung transplant recipient to take home.
- Pocket PATH hand-held device (Experimental): Participants in the intervention group will be trained to use a hand-held device with custom programs as a means of supporting, tracking, and interpreting discharge activities in addition to the standard paper-tracking methods.
  Interventions: Behavioral: Pocket PATH (Personal Assistant for Tracking Health)

INTERVENTIONS:
Behavioral: Pocket PATH (Personal Assistant for Tracking Health) — Participants in the intervention group will be trained to use a hand-held device with custom programs as a means of supporting, tracking, and interpreting discharge activities in addition to the standard paper-tracking methods.
  Arms: Pocket PATH hand-held device

SUMMARY:
The purpose of this randomized controlled trial is to test the efficacy of a novel intervention, Pocket PATH (Personal Assistant for Tracking Health) for promoting self-care agency, self-care behaviors, and transplant-related health.

DETAILED DESCRIPTION:
Lung transplant recipients (LTR) experience more transplant-related complications, higher health resource utilization, and higher mortality than recipients of other solid organs. Prevention and detection of early complications is known to reduce the likelihood of future impairments in lung function and, therefore, morbidity and mortality. Despite the scarce donor organs and financial resources expended to support individuals throughout the lung transplant experience, no randomized controlled trials (RCT) have tested interventions designed to promote self-care behaviors with the aim of improving transplant-related health after lung transplant. The purpose of this RCT is to compare the efficacy of a novel behavioral intervention, Pocket PATH (Personal Assistant for Tracking Health) for promoting self-care and improving health outcomes relative to standard care after lung transplantation. Pocket PATH provides LTR a hand-held device with customized data recording, trending, and decision-support programs to promote their self-care behaviors. Based on the promising results from our early trials, a full-scale RCT has been designed to rigorously test the efficacy of Pocket PATH in promoting self-care agency, self-care behaviors, and hence improving transplant-related health. A sample of 214 LTR who survive the immediate intensive care unit recovery period will be randomly assigned to either the intervention group, who will be instructed to use the Pocket Path device and its programs designed for self-monitoring, adhering to the regimen, and communicating condition changes to the transplant team, or the control group who will receive standard instructions regarding the post-transplant regimen (including health monitoring). Information will be collected from participants at baseline and 1 week, 2, 6, and 12 months after discharge from the hospital following lung transplantation. Longitudinal, repeated-measures models with planned comparisons will be used to test the hypotheses for the primary aims. It is hypothesized that subjects in the Pocket PATH group will develop higher levels of self-care agency and perform self-care behaviors more often than subjects in the control group and, therefore, will experience fewer transplant-related complications, re-hospitalizations, and better health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* a recipient of a lung transplant
* 18 years of age or older
* stable enough to be transferred from the CTICU to the acute unit
* not been discharged from initial transplant hospitalization
* able to read and speak English

Exclusion Criteria:

* a recipient of any prior transplant
* a condition that precludes discharge from the hospital
* limited involvement in post-transplant care is anticipated (e.g., plan to discharge to skilled nursing facility)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Self-care agency and self-care behaviors (performing of self-monitoring, adhering to the medical regimen, communicating with the transplant team) | 1 year post-discharge

SECONDARY OUTCOMES:
Transplant-related health | 1 year post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Annette DeVito Dabbs, PhD, RN, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] DeVito Dabbs A, Song MK, Myers B, Hawkins RP, Aubrecht J, Begey A, Connolly M, Li R, Pilewski JM, Bermudez CA, Dew MA. Clinical trials of health information technology interventions intended for patient use: unique issues and considerations. Clin Trials. 2013;10(6):896-906. doi: 10.1177/1740774513493149. Epub 2013 Jul 18. PMID 23867222
- [Background] Kovach KA, Aubrecht JA, Dew MA, Myers B, Dabbs AD. Data safety and monitoring for research involving remote health monitoring. Telemed J E Health. 2011 Sep;17(7):574-9. doi: 10.1089/tmj.2010.0219. Epub 2011 Jul 12. PMID 21749259
- [Background] Devito Dabbs A, Song MK, Hawkins R, Aubrecht J, Kovach K, Terhorst L, Connolly M, McNulty M, Callan J. An intervention fidelity framework for technology-based behavioral interventions. Nurs Res. 2011 Sep-Oct;60(5):340-7. doi: 10.1097/NNR.0b013e31822cc87d. PMID 21878796
- [Result] DeVito Dabbs A, Song MK, Myers BA, Li R, Hawkins RP, Pilewski JM, Bermudez CA, Aubrecht J, Begey A, Connolly M, Alrawashdeh M, Dew MA. A Randomized Controlled Trial of a Mobile Health Intervention to Promote Self-Management After Lung Transplantation. Am J Transplant. 2016 Jul;16(7):2172-80. doi: 10.1111/ajt.13701. Epub 2016 Mar 14. PMID 26729617
- [Result] Rosenberger EM, DeVito Dabbs AJ, DiMartini AF, Landsittel DP, Pilewski JM, Dew MA. Long-Term Follow-up of a Randomized Controlled Trial Evaluating a Mobile Health Intervention for Self-Management in Lung Transplant Recipients. Am J Transplant. 2017 May;17(5):1286-1293. doi: 10.1111/ajt.14062. Epub 2016 Oct 31. PMID 27664940
- [Result] DeVito Dabbs A, Terhorst L, Song MK, Shellmer DA, Aubrecht J, Connolly M, Dew MA. Quality of recipient-caregiver relationship and psychological distress are correlates of self-care agency after lung transplantation. Clin Transplant. 2013 Jan-Feb;27(1):113-20. doi: 10.1111/ctr.12017. Epub 2012 Sep 24. PMID 23004565
- [Result] Zaldonis J, Alrawashdeh M, Atman KS, Fatigati A, Dabbs AD, Bermudez CA. Predictors and influence of goal orientation on self-management and health-related quality of life after lung transplant. Prog Transplant. 2015 Sep;25(3):230-42. doi: 10.7182/pit2015189. PMID 26308782
- [Result] Fatigati A, Alrawashdeh M, Zaldonis J, Dabbs AD. Patterns and Predictors of Sleep Quality Within the First Year After Lung Transplantation. Prog Transplant. 2016 Mar;26(1):62-9. doi: 10.1177/1526924816632123. PMID 27136251
- [Result] Jiang Y, Sereika SM, DeVito Dabbs A, Handler SM, Schlenk EA. Using mobile health technology to deliver decision support for self-monitoring after lung transplantation. Int J Med Inform. 2016 Oct;94:164-71. doi: 10.1016/j.ijmedinf.2016.07.012. Epub 2016 Jul 19. PMID 27573324
- [Result] Jiang Y, Sereika SM, Dabbs AD, Handler SM, Schlenk EA. Acceptance and Use of Mobile Technology for Health Self-Monitoring in Lung Transplant Recipients during the First Year Post-Transplantation. Appl Clin Inform. 2016 Jun 1;7(2):430-45. doi: 10.4338/ACI-2015-12-RA-0170. eCollection 2016. PMID 27437052
- [Result] Alrawashdeh M, Zomak R, Dew MA, Sereika S, Song MK, Pilewski JM, DeVito Dabbs A. Pattern and Predictors of Hospital Readmission During the First Year After Lung Transplantation. Am J Transplant. 2017 May;17(5):1325-1333. doi: 10.1111/ajt.14064. Epub 2016 Oct 27. PMID 27676226
- [Result] Hu L, Lingler JH, DeVito Dabbs A, Dew MA, Sereika SM. Trajectories of self-care agency and associated factors in lung transplant recipients over the first 12 months following transplantation. Clin Transplant. 2017 Sep;31(9):10.1111/ctr.13030. doi: 10.1111/ctr.13030. Epub 2017 Jul 13. PMID 28609813
- [Result] Hu L, DeVito Dabbs A, Dew MA, Sereika SM, Lingler JH. Patterns and correlates of adherence to self-monitoring in lung transplant recipients during the first 12 months after discharge from transplant. Clin Transplant. 2017 Aug;31(8):10.1111/ctr.13014. doi: 10.1111/ctr.13014. Epub 2017 Jun 11. PMID 28517112
- [Result] Geramita EM, DeVito Dabbs AJ, DiMartini AF, Pilewski JM, Switzer GE, Posluszny DM, Myaskovsky L, Dew MA. Impact of a Mobile Health Intervention on Long-term Nonadherence After Lung Transplantation: Follow-up After a Randomized Controlled Trial. Transplantation. 2020 Mar;104(3):640-651. doi: 10.1097/TP.0000000000002872. PMID 31335759
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- See also: PubMed ID: 26729617 (Abstract) — http://www.ncbi.nlm.nih.gov/pubmed/26729617
- See also: PubMEd ID: 27664940 (Abstract) — https://pubmed.ncbi.nlm.nih.gov/27664940/
- See also: PubMed ID: 23004565 (Abstract) — https://pubmed.ncbi.nlm.nih.gov/23004565/
- See also: PubMed ID: 23867222 (Abstract) — http://pubmed.ncbi.nlm.nih.gov/23867222
- See also: PubMed ID: 26308782 (Abstract) — http://pubmed.ncbi.nlm.nih.gov/26308782
- See also: PubMed ID: 27136251 (Abstract) — http://pubmed.ncbi.nlm.nih.gov/27136251
- See also: Pub Med ID: 27573324 (Abstract) — https://pubmed.ncbi.nlm.nih.gov/27573324
- See also: PubMed ID: 27437052 (Abstract) — http://pubmed.ncbi.nlm.nih.gov/27437052
- See also: PubMed ID: 27676226 (Abstract) — http://pubmed.ncbi.nlm.nih.gov/27676226
- See also: PubMed ID: 28609813 (Abstract) — http://pubmed.ncbi.nlm.nih.gov/28609813
- See also: PubMed ID: 28517112 (Abstract) — http://pubmed.ncbi.nlm.nih.gov/28517112
- See also: PubMed ID: 31335759 (Abstract) — http://pubmed.ncbi.nlm.nih.gov/31335759
- See also: PubMed ID: 21749259 (Abstract) — http://pubmed.ncbi.nlm.nih.gov/21749259
- See also: Pub Med ID: 21878796 — http://pubmed.ncbi.nlm.nih.gov/21878796